CLINICAL TRIAL: NCT03733678
Title: A Sequential and Adaptive Experiment to Increase the Uptake of Long-acting Reversible Contraceptives in Cameroon
Brief Title: A Randomized-Controlled Trial to Increase the Uptake of LARCs in Cameroon
Acronym: HGOPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Collaborators: Stanford University (Other); George Washington University (Other); University of Exeter (Other); University of California, San Diego (Other); Yaounde Gynecology, Obstetrics and Pediatrics Hospital (Unknown)
Responsible Party: Principal Investigator, Berk Ozler, Principal Investigator, World Bank
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: LARCs-2018
Record Dates: First submitted 2018-10-31; First posted 2018-11-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Contraception; Contraception Behavior; Contraceptive Usage; Contraceptive Method Switching
Keywords: adolescent sexual and reproductive health, maternal mortality, teen pregnancy, LARCs, family planning counseling
MeSH Terms: conditions — Contraception Behavior; Maternal Death

STUDY DESIGN:
Intervention Model Description: The study independently experiments with two aspects of the health provider-client relationship:
  1. First, a tablet-based counseling app that is used by the provider gives random discounts to clients - separately for LARCs and SARCs.
  2. Second, the tablet-based app presents recommendations to the client sequentially (i.e. the top-ranked method, followed by the next one if that recommendation is declined by the client, etc.) vs. simultaneously (i.e. presenting the top recommendations to the client all at once and asking her to choose which one to discuss further).
Who Masked: Participant
Masking Description: Participants are masked in some interventions related to the workings of the tablet-based decision-support tool, but not to the price discounts they receive for the contraceptive methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (20):
- Free SARC, Free LARC, Recommendation (Experimental): Free SARC, Free LARC, Sequential recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs
- Free SARC, LARC=500, Recommendation (Experimental): Free SARC, LARC=500 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs
- Free SARC, LARC=1000, Recommendation (Experimental): Free SARC, LARC=1000 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs
- Free SARC, LARC=2140, Recommendation (Experimental): Free SARC, LARC=2140 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs
- Free SARC, LARC=5000, Recommendation (Experimental): Free SARC, LARC=5000 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for SARCs
- Regular SARC, Free LARC, Recommendation (Experimental): Regular price SARC, Free LARC, Sequential recommendation
  Interventions: Behavioral: Price discounts for LARCs
- Regular SARC, LARC=500, Recommendation (Experimental): Regular price SARC, LARC=500 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for LARCs
- Regular SARC, LARC=1000, Recommendation (Experimental): Regular price SARC, LARC=1000 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for LARCs
- Regular SARC, LARC=2140, Recommendation (Experimental): Regular price SARC, LARC=2140 CFA, Sequential recommendation
  Interventions: Behavioral: Price discounts for LARCs
- Regular SARC, LARC=5000, Recommendation (No Intervention): Regular price SARC, LARC=5000 CFA, Sequential recommendation
- Free SARC, Free LARC, No Recommendation (Experimental): Free SARC, Free LARC, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Free SARC, LARC=500, No Recommendation (Experimental): Free SARC, LARC=500 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Free SARC, LARC=1000, No Recommendation (Experimental): Free SARC, LARC=1000 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Free SARC, LARC=2140, No Recommendation (Experimental): Free SARC, LARC=2140 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Free SARC, LARC=5000, No Recommendation (Experimental): Free SARC, LARC=5000 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for SARCs; Behavioral: Sequential vs. simultaneous recommendations
- Regular SARC, Free LARC, No Recommendation (Experimental): Regular Price SARC, Free LARC, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Regular SARC, LARC=500, No Recommendation (Experimental): Regular Price SARC, LARC=500 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Regular SARC, LARC=1000, No Recommendation (Experimental): Regular Price SARC, LARC=1000 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Regular SARC, LARC=2140, No Recommendation (Experimental): Regular Price SARC, LARC=2140 CFA, Simultaneous recommendation
  Interventions: Behavioral: Price discounts for LARCs; Behavioral: Sequential vs. simultaneous recommendations
- Regular SARC, LARC=5000, No Recommendation (Experimental): Regular Price SARC, LARC=5000 CFA, Simultaneous recommendation
  Interventions: Behavioral: Sequential vs. simultaneous recommendations

INTERVENTIONS:
Behavioral: Price discounts for SARCs — SARCs are offered free to the client
  Arms: Free SARC, Free LARC, No Recommendation; Free SARC, Free LARC, Recommendation; Free SARC, LARC=1000, No Recommendation; Free SARC, LARC=1000, Recommendation; Free SARC, LARC=2140, No Recommendation; Free SARC, LARC=2140, Recommendation; Free SARC, LARC=500, No Recommendation; Free SARC, LARC=500, Recommendation; Free SARC, LARC=5000, No Recommendation; Free SARC, LARC=5000, Recommendation
Behavioral: Price discounts for LARCs — LARCs are offered at lower prices to the client
  Arms: Free SARC, Free LARC, No Recommendation; Free SARC, Free LARC, Recommendation; Free SARC, LARC=1000, No Recommendation; Free SARC, LARC=1000, Recommendation; Free SARC, LARC=2140, No Recommendation; Free SARC, LARC=2140, Recommendation; Free SARC, LARC=500, No Recommendation; Free SARC, LARC=500, Recommendation; Regular SARC, Free LARC, No Recommendation; Regular SARC, Free LARC, Recommendation; Regular SARC, LARC=1000, No Recommendation; Regular SARC, LARC=1000, Recommendation; Regular SARC, LARC=2140, No Recommendation; Regular SARC, LARC=2140, Recommendation; Regular SARC, LARC=500, No Recommendation; Regular SARC, LARC=500, Recommendation
Behavioral: Sequential vs. simultaneous recommendations — Top ranked methods are presented to the client sequentially or simultaneously
  Arms: Free SARC, Free LARC, No Recommendation; Free SARC, LARC=1000, No Recommendation; Free SARC, LARC=2140, No Recommendation; Free SARC, LARC=500, No Recommendation; Free SARC, LARC=5000, No Recommendation; Regular SARC, Free LARC, No Recommendation; Regular SARC, LARC=1000, No Recommendation; Regular SARC, LARC=2140, No Recommendation; Regular SARC, LARC=500, No Recommendation; Regular SARC, LARC=5000, No Recommendation

SUMMARY:
Cameroon exhibits a high and non-decreasing level of maternal mortality (roughly 600 per 100,000 live births), partially related to its relatively high total fertility rate (roughly 4.6). Survey evidence furthermore suggests that a significant fraction of these pregnancies is unwanted or considered mistimed by the mother, especially among females aged 15-19. Despite this, the rate of utilization of family planning (FP) is low: e.g. only 48% of sexually active unmarried women use any form of (modern) contraception, or MC, and even then, it is primarily condoms. The use of LARCs (long-acting reversible contraceptives, i.e. the IUD and implant) is less than 1% according to the most recent Demographic Health Survey.

The study investigators propose to use an integrated behavioral science approach to increase the take-up of both SARCs (short-acting reversible contraceptives, i.e. the pill and injectable) and especially LARCs among reproductive-age females in Cameroon, including adolescents who may be unmarried and/or nulliparous. In addition to decreasing maternal mortality and undesired pregnancies, indirect effects for the community will include: increased welfare from reduced side effects that arise due to current one-size-fits-all FP counseling; healthier children due to improved birth spacing; and increased human capital formation both for children and for young (often school-aged) potential mothers.

The study investigators propose to conduct the study at HGOPY for a duration of 12 months. The study investigators will provide tablets to each of five nurses that conduct FP counseling to participants at the hospital. The tablets contain a counseling "app" (or decision-support tool or a job-aid) that was jointly developed by professionals from HGOPY, the World Bank, and the Ministry of Health. The study investigators propose an individually-randomized experiment, where the participants will be offered randomly varying discounts for the modern contraceptive methods they wish to adopt. The study investigators also propose to experiment with certain aspects of the "app" to improve its effectiveness - both for the participant and for the nurse. More details on the experimental design are provided below.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 10-49
* Presenting at HGOPY seeking FP counseling/services
* HGOPY clients referred to the family planning unit for consultation

Exclusion Criteria:

* No exclusion criteria

Ages: 10 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2500 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The client adopted a LARC | 1-day
  using data from the counseling sessions
The client adopted a modern contraceptive method (LARC or SARC) | 1-day
  using data from the counseling sessions

SECONDARY OUTCOMES:
Was the client treated with respect by the provider during the counseling session? | 2-weeks
  Self-reported indicator variable using follow-up surveys two weeks after counseling session
Did the client trust the provider during the counseling session? | 2-weeks
  Self-reported indicator variable using follow-up surveys two weeks after counseling session
Did the health provider give information about contraceptive methods that was easy to understand during the counseling session? | 2-weeks
  Self-reported indicator variable using follow-up surveys two weeks after counseling session
Client satisfaction with adopted contraceptive method | 2-week and 16-week measurements
  using 2-week and 16-week follow-up surveys
Discontinuation of adopted contraceptive method | 2-week, 16-week, and 52-week measurements
  using 2-week, 16-week, and 52-week follow-up surveys
Percentage of participants with unintended pregnancy within the time frame | 16-week and 52-week measurements
  using 16-week and 52-week follow-up surveys

CONTACTS AND LOCATIONS:
Overall Officials: Berk Ozler, PhD, Principal Investigator — World Bank
Locations (1):
- Hôpital gynéco-obstétrique et pédiatrique de Yaoundé (HGOPY), Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided
We will likely share de-identified anonymous participant data publicly after the trial ends and our analyses are completed.